CLINICAL TRIAL: NCT05151718
Title: Ependymomics: Multiomic Approach to Radioresistance of Ependymomas in Children and Adolescents
Brief Title: Multiomic Approach to Radioresistance of Ependymomas in Children and Adolescents
Acronym: EPENDYMOMICS
Status: Recruiting | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre Leon Berard (Other); Assistance Publique Hopitaux De Marseille (Other); Centre Hospitalier St Anne (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 21 HLTETE 01
Record Dates: First submitted 2021-12-08; First posted 2021-12-09 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Ependymoma of Brain; Pediatric Solid Tumor
Keywords: childhood ependymoma; radio-resistance; radiogenomic signature
MeSH Terms: conditions — Familial ependymoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE sample of each patient tumor is included in the PEPPI cohort to Marseille is stored in the AP-HM tumor bank (AP-HM CRB-TBM (Centre de Ressources Biologiques - Tumorothèque et Banque de Muscle - CRB BB-0033-00097) headed by Prof D. Figarella-Branger, certified Afnor 96900 and ISO 9001 (AC-2018-3105) until use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Treatment of childhood ependymoma, the second most frequent pediatric brain tumor, is based on surgery and radiation therapy. However, 50% relapse, mainly locally. Progress in imaging, molecular biology and radiotherapy ballistics has led us to propose the EPENDYMOMICS project, a multi-omics approach using artificial intelligence to detect the predictive characteristics of relapse, and to define innovative radiotherapy targets using multimodal imaging. We previously reported that the relapse sites are mainly located in the high-dose radiotherapy zone and that there appear to be prognostic factors for relapse based on anatomical and functional MRI abnormalities by diffusion and perfusion. In addition, recent studies in molecular biology have identified significant prognostic factors. The challenge now is to use and correlate all these findings in larger cohorts to tackle the radio-resistance of this disease.

Our objective is to collate in a single database called NETSPARE (Network to Structure and Share Pediatric data to Accelerate Research on Ependymoma) the clinical, histological, biological, imaging and radiotherapy data from two consecutive studies that included 370 children and adolescents with ependymoma since 2000 in France. The EPENDYMOMICS project will comprise a clinical research team, three imaging research teams, two histopathology teams, and a biostatistics team working on NETSPARE. Our goal is to obtain a radiogenomic signature of our data, which will be validated with the English external cohort of 200 patients that is currently being analyzed. The perspective is to optimize the indications and volumes of irradiation that could in the future be used in a European translational research trial to tackle radioresistance.

DETAILED DESCRIPTION:
The resistance to treatment prompted us to perform the national PEPPI study (Pediatric Ependymoma Photons Protons and Imaging). PEPPI collated clinical, imaging and dosimetry data from children with intracranial ependymoma treated in France between 2000 and 2013. Since then, patients are treated in the current prospective SIOP II Ependymoma program. Our clinical results confirmed the classical clinical prognostic factors including radiotherapy dose, and we showed that imaging biomarkers from T2/FLAIR, perfusion and diffusion MRI were novel prognostic factors. We reported that relapse after RT occurs mainly locally within the high-dose region. The prognostic value of dose and the high rate of relapse with standard dose prompted us to perform an in silico dosimetry study of dose escalation comparing photons and protons, confirming the feasibility of this approach. In PEPPI series, the prediction of the site of relapse with advanced MR imaging was not possible due to small sample of imaging data and the recent biomolecular classification was not available. Recently, DNA methylation profiling provided a novel classification of ependymoma in molecular subgroups harbouring a strong prognostic value.

EPENDYMOMICS project aims to determine the prognostic role of multimodal imaging, to identify radioresistant clusters predictive of relapse and to analyze the link between radiomics features and genomic markers, hence leading to a radiogenomics study. It will build on a database with a larger number of patients called NETSPARE (Network to Structure and Share Pediatric data to Accelerate Research on Ependymoma) to develop a radiomics approach, i.e. predict clinical endpoints by relying on quantitative features extracted from medical images using either handcrafted or automated features extraction algorithms. These features will be exploited and combined with other available variables (clinical, genetic, etc.) as improved decision support.

1. Data collection MRI: Diagnostic, FU until relapse (DICOM format)

   - Sequences: T1W, T2W, FLAIR, T1W with & without contrast enhancement, diffusion-weighted imaging (DWI), perfusion-weighted imaging (PWI) Radiotherapy: CT scan, RTDOSE, RTSS, RTPLAN (DICOM RT format) Clinical: Age, surgery, chemotherapy, doses, late effects, relapse date Histology: Hematoxylin and Eosin (H&E)-stained histopathology slides Molecular Biology: Methylation groups RELA, YAP, PFA, and PFB
2. Data quality check and delineation of volume of interest to curate data before post-processing and analysis.

   To ensure preliminary robust image segmentation the Radiotherapy Structure Set will be checked for each patient. The referring radiologist will confirm all imaging changes after RT. An expert radiation oncologist will segment volumes of post-treatment abnormalities in T1WI post contrast, in T2W/FLAIR imaging, as well as site of relapse and missing OARs.
3. Imaging data post-processing and analysis of changes after radiotherapy We will process the DWI and PWI with the Olea Sphere®3.0 software, a post-processing solution for MRI and CT scanners. We will extract and generate Apparent Diffusion Coefficient maps from DWI data calculated on a voxel-by-voxel basis and relative cerebral blood volume maps calculated from PWI data with an oscillation-index singular value decomposition routine and correction for T1-weighted leakage effects.

   All the MRI data will be strictly co-registered with the T1WI-PC and planning CT.
4. Radiomics harmonization We will perform the increase of the level of harmonization of images and/or extracted features on highly heterogeneous dataset due to its multiple sources.

   We will develop a GAN-based framework, translating heterogeneous images to match the properties of a standard dataset, such as a template reference image, or alternatively, one set of images chosen as a reference. We need to determine the relevant properties within images (local or global metrics, texture, edges, contrast, signal-to-noise ratio, etc.) and to ensure the ability of the framework to harmonize images without losing their clinically relevant informative and content.

   In the features space, numerous statistical approaches can be applied, such as normalization or batch effect compensation. ComBat has been shown to outperform other similar approaches and we will rely on Monte Carlo estimation for small samples. We will investigate the combination of the batch-correction methods with unsupervised clustering to deal with data presenting very high heterogeneity and a very small number of samples per batch.

   It might be beneficial and complementary to combine image-based and feature-based harmonization methodologies for improving the results of multicenter radiomics studies. We will evaluate the potential added benefit of both previously developed approaches in improving the results. The goal of this task will be to establish whether the first or the second approach (or the combination of both) is the most efficient, taking into account not only the absolute improvement observed in the results, but also the computing time and effort required to implement each approach in practice.
5. Biomolecular analysis Biological resources from PEPPI and SIOPII ependymoma cohorts of patients will be included. First, the diagnosis of intracranial ependymomas will be confirmed and then pathological features will be investigated.

   WHO 2020 classification of ependymomas: the cIMPACT-NOW (Consortium to Inform Molecular and Practical Approaches to CNS Tumor Taxonomy - Not Official WHO) decided to classify ependymomas according to location and the underlying genetic alteration. The current WHO classification is under revision.

   Biological studies required to classify intracranial ependymoma of the project:

   Immunohistochemistry: p65-RelA, H3K27Me3. FISH analysis (classification and Copy Number Variations). DNA-methylation profiling. RNAseq analysis.
6. Deep learning (DL) for molecular biomarkers of ependymoma For this purpose, the Zimmer team has designed and trained deep convolutional neural networks based on the Inception V3 architecture to distinguish ependymoma from glioma grades III and IV. Preliminary results based on an imaging data set indicate a high accuracy of discrimination and suggest the possibility to predict clinically relevant mutations from H&E images alone (manuscript in preparation).

   We will extend these DL approaches to predict resistance to therapy and metastasis. This will be done by using the histopathology images alone either as input or in combination with classifications based on molecular assays. At a technical level, we will use state-of-the-art deep neural network architectures based on convolutional layers and skip connections. To compensate for the moderate size of the training data set, we will make heavy use of transfer learning. Here, we will make specific use of the TGCA database, which contains images from very different cancers such as breast cancer, and adapt successful models by retraining on a subset of the ependymoma data acquired in this study. We also will adopt multi-scale image representations for a better exploitation of the image information at cellular and tissue levels, use H&E specific color normalization and methods for automated elimination of regions subject to imaging artefacts. We also will incorporate the developed methods in Imjoy. By decoupling the graphical user interface from the computational back end, it enables users to access high-end computing capabilities from any workstation or laptop.
7. Statistical analysis Several signatures will be developed and validated : a radiomic signature (RAD-Score), a radiomic and clinical signature (RADClin-Score), a molecular signature (MOL-score) and a global signature (Radiomic, Molecular and clinical signature).

   * RAD-Score associated with progression-free survival (PFS). To avoid biases, NETSPARE built from retrospective multicenter study including independent cohorts is a training cohort. The validation cohort to test the performance of the radiomic signature corresponds to the UK cohort of SIOP II Program (n=220). This division allows external validation.

Training Cohort: the median PFS is estimated to be 5 years in literature. This corresponds to a 3.5-year PFS of 62%. With 370 patients and a median follow-up of 3.5 years, we expect at least 120 events. According to the rule of thumb recommending 10 events per variable of interest, a multiparametric model combining 10 variables may be trained. An alternative modeling strategy based on a penalized approach will be used to study the association between imaging parameters and PFS. As imaging biomarker data far exceeds sample size and are intercorrelated, penalized methods (previously used in different situations with spatial data) will be used for the regularization and selection of variables, by encouraging the grouping effect and select explanatory variables.

Validation cohort: 66 events are expected. With this number of events, it is possible to detect with 80% power a hazard ratio of 0.5 between the low- and high-risk group (Logrank test two-sided 0.05).

Demographic data: Continuous variables will be summarized by cohort using median, minimum, maximum and number of available observations. Qualitative variables will be summarized using counts, percentages and number of missing data. Comparison between cohort will be performed using the chi-square test (or Fisher exact test if applicable) for qualitative variables and the Mann-Whitney test for quantitative variables.

- Radiomics signature development and validation: To study the association between imaging features and PFS, we will use an alternative modeling strategy based on the penalized Cox regression model. Elastic Net method encourages grouping effect and selects explanatory variables. We will perform a 10-fold cross-validation to select the best penalty parameter lambda. The mixing parameter α, other parameter of the Elastic net method, will be set to a default value of 0.5. The regression coefficients associated with each state of the different variables will be used to determine the RAD score. As the outcome is time-dependent, the risk score will be dichotomized using a time-dependent ROC curve to obtain a classifier (risk groups: poor vs intermediate vs good prognosis). The optimal threshold has been determined to obtain at 3 years a sensitivity of at least 80% and the best specificity.

An interval validation will be performed using a leave k-out cross-validation. We will then apply the RAD-score signature to the validation cohort. Performances of the score will be evaluated using different criteria: monotonicity of the prognostic stratification assessed using Kaplan-Meier survival curves and Hazard Ratio (HR) estimation, discrimination evaluated by Harrell's C-Index and the D statistics, quality of the model and the proportion of explained variation estimated by the Akaike Information Criterion (AIC) and the RD² statistic, respectively. The ability of prognostic score to identify patients at high risk of relapse during the first 3 years will be evaluated by determining the sensitivity, specificity and predictive value using a time-dependent ROC curve.

- RADClin-Score development and validation: To incorporate clinical and imaging informations, we will combine both low-dimensional clinical and high-dimensional imaging data in a global prediction model. First, we will completely ignore the imaging features. A Cox model will be fitted to identify clinical covariates associated with PFS. We will build a clinical linear predictor using a regression coefficient. Next, we will use Elastic Net with the clinical linear predictor in offset to identify imaging features. Finally, we will compute the RADClin-Score using a regression coefficient. We will plot a Venn diagram to compare feature selection with the RADClin-Score and the RAD-Score. We will compare the model using the different criteria previously presented.

ELIGIBILITY:
Inclusion Criteria:

* children with intracranial ependymoma
* treated
* included in PEPPI study, pediaRT or in SIOP II Ependymoma french program

Exclusion Criteria:

* NA

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with intracranial ependymoma treated in France since 2000 (included in PEPPI study between 2000 and 2013 and in pediaRT and french SIOP II programme since 2013)
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Definition of radiogenomics signatures that are predictive of patient outcome | 30 months
  The primary endpoint is progression-free survival (PFS), i.e. the time from diagnosis to progression or death from any cause. Patients alive at last follow-up are censored at this date.

SECONDARY OUTCOMES:
Definition of new RT target volumes based on radiomic features and to choose their indications based on biomolecular prognostic factors | 30 months
  Several indexes will be used to evaluate discriminant capacity: Harrell's C-Index and the D statistics, Akaike Information Criterion (AIC) and the RD² statistic
To predict resistance to therapy by using the histological data in digital format and the biomolecular data for analysis by methods based on artificial deep neural networks . | 30 months
  Several indexes will be used to evaluate discriminant capacity: Harrell's C-Index and the D statistics, Akaike Information Criterion (AIC) and the RD² statistic

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claudius Regaud, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tensaouti F, Ducassou A, Chaltiel L, Bolle S, Muracciole X, Coche-Dequeant B, Alapetite C, Bernier V, Claude L, Supiot S, Huchet A, Kerr C, le Prise E, Laprie A; radiotherapy committee of the French Society for Childhood Cancer (SFCE). Patterns of failure after radiotherapy for pediatric patients with intracranial ependymoma. Radiother Oncol. 2017 Mar;122(3):362-367. doi: 10.1016/j.radonc.2016.12.025. Epub 2017 Jan 12. PMID 28089483
- [Background] Ducassou A, Padovani L, Chaltiel L, Bolle S, Habrand JL, Claude L, Carrie C, Muracciole X, Coche-Dequeant B, Alapetite C, Supiot S, Demoor-Goldschmidt C, Bernier-Chastagner V, Huchet A, Leseur J, Le Prise E, Kerr C, Truc G, Nguyen TD, Bertozzi AI, Frappaz D, Boetto S, Sevely A, Tensaouti F, Laprie A; Pediatric French Radiation Oncologist Group (GFRP) and the French Society of Children With Cancer (SFCE). Pediatric Localized Intracranial Ependymomas: A Multicenter Analysis of the Societe Francaise de lutte contre les Cancers de l'Enfant (SFCE) from 2000 to 2013. Int J Radiat Oncol Biol Phys. 2018 Sep 1;102(1):166-173. doi: 10.1016/j.ijrobp.2018.05.036. Epub 2018 May 24. PMID 30102193
- [Background] Tensaouti F, Ducassou A, Chaltiel L, Sevely A, Bolle S, Muracciole X, Coche-Dequant B, Alapetite C, Supiot S, Huchet A, Bernier V, Claude L, Bertozzi-Salamon AI, Liceaga S, Lotterie JA, Peran P, Payoux P, Laprie A; radiotherapy committee of the French Society for Childhood Cancer (SFCE). Prognostic and predictive values of diffusion and perfusion MRI in paediatric intracranial ependymomas in a large national study. Br J Radiol. 2016 Oct;89(1066):20160537. doi: 10.1259/bjr.20160537. Epub 2016 Aug 23. PMID 27550423
- [Background] Tensaouti F, Ducassou A, Chaltiel L, Sevely A, Bolle S, Padovani L, Jouin A, Alapetite C, Supiot S, Huchet A, Bernier V, Claude L, Kerr C, Le Prise E, Bertozzi-Salamon AI, Liceaga S, Lotterie JA, Peran P, Laprie A; French Society for Childhood Cancer (SFCE). Imaging biomarkers of outcome after radiotherapy for pediatric ependymoma. Radiother Oncol. 2018 Apr;127(1):103-107. doi: 10.1016/j.radonc.2018.02.008. Epub 2018 Mar 2. PMID 29500084
- [Background] Tensaouti F, Ducassou A, Chaltiel L, Bolle S, Habrand JL, Alapetite C, Coche-Dequeant B, Bernier V, Claude L, Carrie C, Padovani L, Muracciole X, Supiot S, Huchet A, Leseur J, Kerr C, Hangard G, Lisbona A, Goudjil F, Ferrand R, Laprie A. Feasibility of Dose Escalation in Patients With Intracranial Pediatric Ependymoma. Front Oncol. 2019 Jun 21;9:531. doi: 10.3389/fonc.2019.00531. eCollection 2019. PMID 31293971
- [Background] Pajtler KW, Mack SC, Ramaswamy V, Smith CA, Witt H, Smith A, Hansford JR, von Hoff K, Wright KD, Hwang E, Frappaz D, Kanemura Y, Massimino M, Faure-Conter C, Modena P, Tabori U, Warren KE, Holland EC, Ichimura K, Giangaspero F, Castel D, von Deimling A, Kool M, Dirks PB, Grundy RG, Foreman NK, Gajjar A, Korshunov A, Finlay J, Gilbertson RJ, Ellison DW, Aldape KD, Merchant TE, Bouffet E, Pfister SM, Taylor MD. The current consensus on the clinical management of intracranial ependymoma and its distinct molecular variants. Acta Neuropathol. 2017 Jan;133(1):5-12. doi: 10.1007/s00401-016-1643-0. Epub 2016 Nov 17. PMID 27858204
- [Background] Da-Ano R, Visvikis D, Hatt M. Harmonization strategies for multicenter radiomics investigations. Phys Med Biol. 2020 Dec 17;65(24):24TR02. doi: 10.1088/1361-6560/aba798. PMID 32688357
- [Background] Johnson WE, Li C, Rabinovic A. Adjusting batch effects in microarray expression data using empirical Bayes methods. Biostatistics. 2007 Jan;8(1):118-27. doi: 10.1093/biostatistics/kxj037. Epub 2006 Apr 21. PMID 16632515
- [Background] Chen C, Grennan K, Badner J, Zhang D, Gershon E, Jin L, Liu C. Removing batch effects in analysis of expression microarray data: an evaluation of six batch adjustment methods. PLoS One. 2011 Feb 28;6(2):e17238. doi: 10.1371/journal.pone.0017238. PMID 21386892
- [Background] Da-Ano R, Masson I, Lucia F, Dore M, Robin P, Alfieri J, Rousseau C, Mervoyer A, Reinhold C, Castelli J, De Crevoisier R, Ramee JF, Pradier O, Schick U, Visvikis D, Hatt M. Performance comparison of modified ComBat for harmonization of radiomic features for multicenter studies. Sci Rep. 2020 Jun 24;10(1):10248. doi: 10.1038/s41598-020-66110-w. PMID 32581221
- [Background] Louis DN, Wesseling P, Aldape K, Brat DJ, Capper D, Cree IA, Eberhart C, Figarella-Branger D, Fouladi M, Fuller GN, Giannini C, Haberler C, Hawkins C, Komori T, Kros JM, Ng HK, Orr BA, Park SH, Paulus W, Perry A, Pietsch T, Reifenberger G, Rosenblum M, Rous B, Sahm F, Sarkar C, Solomon DA, Tabori U, van den Bent MJ, von Deimling A, Weller M, White VA, Ellison DW. cIMPACT-NOW update 6: new entity and diagnostic principle recommendations of the cIMPACT-Utrecht meeting on future CNS tumor classification and grading. Brain Pathol. 2020 Jul;30(4):844-856. doi: 10.1111/bpa.12832. Epub 2020 Apr 19. PMID 32307792
- [Background] Louis DN, Perry A, Reifenberger G, von Deimling A, Figarella-Branger D, Cavenee WK, Ohgaki H, Wiestler OD, Kleihues P, Ellison DW. The 2016 World Health Organization Classification of Tumors of the Central Nervous System: a summary. Acta Neuropathol. 2016 Jun;131(6):803-20. doi: 10.1007/s00401-016-1545-1. Epub 2016 May 9. PMID 27157931
- [Background] Parker M, Mohankumar KM, Punchihewa C, Weinlich R, Dalton JD, Li Y, Lee R, Tatevossian RG, Phoenix TN, Thiruvenkatam R, White E, Tang B, Orisme W, Gupta K, Rusch M, Chen X, Li Y, Nagahawhatte P, Hedlund E, Finkelstein D, Wu G, Shurtleff S, Easton J, Boggs K, Yergeau D, Vadodaria B, Mulder HL, Becksfort J, Gupta P, Huether R, Ma J, Song G, Gajjar A, Merchant T, Boop F, Smith AA, Ding L, Lu C, Ochoa K, Zhao D, Fulton RS, Fulton LL, Mardis ER, Wilson RK, Downing JR, Green DR, Zhang J, Ellison DW, Gilbertson RJ. C11orf95-RELA fusions drive oncogenic NF-kappaB signalling in ependymoma. Nature. 2014 Feb 27;506(7489):451-5. doi: 10.1038/nature13109. Epub 2014 Feb 19. PMID 24553141
- [Background] Panwalkar P, Clark J, Ramaswamy V, Hawes D, Yang F, Dunham C, Yip S, Hukin J, Sun Y, Schipper MJ, Chavez L, Margol A, Pekmezci M, Chung C, Banda A, Bayliss JM, Curry SJ, Santi M, Rodriguez FJ, Snuderl M, Karajannis MA, Saratsis AM, Horbinski CM, Carret AS, Wilson B, Johnston D, Lafay-Cousin L, Zelcer S, Eisenstat D, Silva M, Scheinemann K, Jabado N, McNeely PD, Kool M, Pfister SM, Taylor MD, Hawkins C, Korshunov A, Judkins AR, Venneti S. Immunohistochemical analysis of H3K27me3 demonstrates global reduction in group-A childhood posterior fossa ependymoma and is a powerful predictor of outcome. Acta Neuropathol. 2017 Nov;134(5):705-714. doi: 10.1007/s00401-017-1752-4. Epub 2017 Jul 21. PMID 28733933
- [Background] Pajtler KW, Witt H, Sill M, Jones DT, Hovestadt V, Kratochwil F, Wani K, Tatevossian R, Punchihewa C, Johann P, Reimand J, Warnatz HJ, Ryzhova M, Mack S, Ramaswamy V, Capper D, Schweizer L, Sieber L, Wittmann A, Huang Z, van Sluis P, Volckmann R, Koster J, Versteeg R, Fults D, Toledano H, Avigad S, Hoffman LM, Donson AM, Foreman N, Hewer E, Zitterbart K, Gilbert M, Armstrong TS, Gupta N, Allen JC, Karajannis MA, Zagzag D, Hasselblatt M, Kulozik AE, Witt O, Collins VP, von Hoff K, Rutkowski S, Pietsch T, Bader G, Yaspo ML, von Deimling A, Lichter P, Taylor MD, Gilbertson R, Ellison DW, Aldape K, Korshunov A, Kool M, Pfister SM. Molecular Classification of Ependymal Tumors across All CNS Compartments, Histopathological Grades, and Age Groups. Cancer Cell. 2015 May 11;27(5):728-43. doi: 10.1016/j.ccell.2015.04.002. PMID 25965575
- [Background] Pajtler KW, Wen J, Sill M, Lin T, Orisme W, Tang B, Hubner JM, Ramaswamy V, Jia S, Dalton JD, Haupfear K, Rogers HA, Punchihewa C, Lee R, Easton J, Wu G, Ritzmann TA, Chapman R, Chavez L, Boop FA, Klimo P, Sabin ND, Ogg R, Mack SC, Freibaum BD, Kim HJ, Witt H, Jones DTW, Vo B, Gajjar A, Pounds S, Onar-Thomas A, Roussel MF, Zhang J, Taylor JP, Merchant TE, Grundy R, Tatevossian RG, Taylor MD, Pfister SM, Korshunov A, Kool M, Ellison DW. Molecular heterogeneity and CXorf67 alterations in posterior fossa group A (PFA) ependymomas. Acta Neuropathol. 2018 Aug;136(2):211-226. doi: 10.1007/s00401-018-1877-0. Epub 2018 Jun 16. PMID 29909548
- [Background] Siegfried A, Rousseau A, Maurage CA, Pericart S, Nicaise Y, Escudie F, Grand D, Delrieu A, Gomez-Brouchet A, Le Guellec S, Franchet C, Boetto S, Vinchon M, Sol JC, Roux FE, Rigau V, Bertozzi AI, Jones DTW, Figarella-Branger D, Uro-Coste E. EWSR1-PATZ1 gene fusion may define a new glioneuronal tumor entity. Brain Pathol. 2019 Jan;29(1):53-62. doi: 10.1111/bpa.12619. Epub 2018 Jul 13. PMID 29679497
- [Background] Siegfried A, Masliah-Planchon J, Roux FE, Larrieu-Ciron D, Pierron G, Nicaise Y, Gambart M, Catalaa I, Pericart S, Dubucs C, Mohand-Oumoussa B, Tirode F, Bourdeaut F, Uro-Coste E. Brain tumor with an ATXN1-NUTM1 fusion gene expands the histologic spectrum of NUTM1-rearranged neoplasia. Acta Neuropathol Commun. 2019 Dec 30;7(1):220. doi: 10.1186/s40478-019-0870-8. No abstract available. PMID 31888756
- [Background] Kermany DS, Goldbaum M, Cai W, Valentim CCS, Liang H, Baxter SL, McKeown A, Yang G, Wu X, Yan F, Dong J, Prasadha MK, Pei J, Ting MYL, Zhu J, Li C, Hewett S, Dong J, Ziyar I, Shi A, Zhang R, Zheng L, Hou R, Shi W, Fu X, Duan Y, Huu VAN, Wen C, Zhang ED, Zhang CL, Li O, Wang X, Singer MA, Sun X, Xu J, Tafreshi A, Lewis MA, Xia H, Zhang K. Identifying Medical Diagnoses and Treatable Diseases by Image-Based Deep Learning. Cell. 2018 Feb 22;172(5):1122-1131.e9. doi: 10.1016/j.cell.2018.02.010. PMID 29474911
- [Background] Coudray N, Ocampo PS, Sakellaropoulos T, Narula N, Snuderl M, Fenyo D, Moreira AL, Razavian N, Tsirigos A. Classification and mutation prediction from non-small cell lung cancer histopathology images using deep learning. Nat Med. 2018 Oct;24(10):1559-1567. doi: 10.1038/s41591-018-0177-5. Epub 2018 Sep 17. PMID 30224757
- [Background] Vahadane A, Peng T, Sethi A, Albarqouni S, Wang L, Baust M, Steiger K, Schlitter AM, Esposito I, Navab N. Structure-Preserving Color Normalization and Sparse Stain Separation for Histological Images. IEEE Trans Med Imaging. 2016 Aug;35(8):1962-71. doi: 10.1109/TMI.2016.2529665. Epub 2016 Apr 27. PMID 27164577
- [Background] Ouyang W, Mueller F, Hjelmare M, Lundberg E, Zimmer C. ImJoy: an open-source computational platform for the deep learning era. Nat Methods. 2019 Dec;16(12):1199-1200. doi: 10.1038/s41592-019-0627-0. No abstract available. PMID 31780825
- [Background] Moons KG, Altman DG, Vergouwe Y, Royston P. Prognosis and prognostic research: application and impact of prognostic models in clinical practice. BMJ. 2009 Jun 4;338:b606. doi: 10.1136/bmj.b606. No abstract available. PMID 19502216
- [Background] Deist TM, Dankers FJWM, Valdes G, Wijsman R, Hsu IC, Oberije C, Lustberg T, van Soest J, Hoebers F, Jochems A, El Naqa I, Wee L, Morin O, Raleigh DR, Bots W, Kaanders JH, Belderbos J, Kwint M, Solberg T, Monshouwer R, Bussink J, Dekker A, Lambin P. Machine learning algorithms for outcome prediction in (chemo)radiotherapy: An empirical comparison of classifiers. Med Phys. 2018 Jul;45(7):3449-3459. doi: 10.1002/mp.12967. Epub 2018 Jun 13. PMID 29763967
- [Background] Cozzi L, Dinapoli N, Fogliata A, Hsu WC, Reggiori G, Lobefalo F, Kirienko M, Sollini M, Franceschini D, Comito T, Franzese C, Scorsetti M, Wang PM. Radiomics based analysis to predict local control and survival in hepatocellular carcinoma patients treated with volumetric modulated arc therapy. BMC Cancer. 2017 Dec 6;17(1):829. doi: 10.1186/s12885-017-3847-7. PMID 29207975
- [Background] Collins GS, Reitsma JB, Altman DG, Moons KG. Transparent reporting of a multivariable prediction model for individual prognosis or diagnosis (TRIPOD): the TRIPOD statement. BMJ. 2015 Jan 7;350:g7594. doi: 10.1136/bmj.g7594. PMID 25569120
- [Background] Royston P, Sauerbrei W. A new measure of prognostic separation in survival data. Stat Med. 2004 Mar 15;23(5):723-48. doi: 10.1002/sim.1621. PMID 14981672
- [Background] Heagerty PJ, Zheng Y. Survival model predictive accuracy and ROC curves. Biometrics. 2005 Mar;61(1):92-105. doi: 10.1111/j.0006-341X.2005.030814.x. PMID 15737082
- [Background] De Bin R, Sauerbrei W, Boulesteix AL. Investigating the prediction ability of survival models based on both clinical and omics data: two case studies. Stat Med. 2014 Dec 30;33(30):5310-29. doi: 10.1002/sim.6246. Epub 2014 Jul 9. PMID 25042390
- [Background] Laprie A, Ken S, Filleron T, Lubrano V, Vieillevigne L, Tensaouti F, Catalaa I, Boetto S, Khalifa J, Attal J, Peyraga G, Gomez-Roca C, Uro-Coste E, Noel G, Truc G, Sunyach MP, Magne N, Charissoux M, Supiot S, Bernier V, Mounier M, Poublanc M, Fabre A, Delord JP, Cohen-Jonathan Moyal E. Dose-painting multicenter phase III trial in newly diagnosed glioblastoma: the SPECTRO-GLIO trial comparing arm A standard radiochemotherapy to arm B radiochemotherapy with simultaneous integrated boost guided by MR spectroscopic imaging. BMC Cancer. 2019 Feb 21;19(1):167. doi: 10.1186/s12885-019-5317-x. PMID 30791889
- [Background] Khalifa J, Tensaouti F, Lotterie JA, Catalaa I, Chaltiel L, Benouaich-Amiel A, Gomez-Roca C, Noel G, Truc G, Peran P, Berry I, Sunyach MP, Charissoux M, Johnson C, Cohen-Jonathan Moyal E, Laprie A. Do perfusion and diffusion MRI predict glioblastoma relapse sites following chemoradiation? J Neurooncol. 2016 Oct;130(1):181-192. doi: 10.1007/s11060-016-2232-8. Epub 2016 Aug 8. PMID 27502603
- [Background] Laprie A, Catalaa I, Cassol E, McKnight TR, Berchery D, Marre D, Bachaud JM, Berry I, Moyal EC. Proton magnetic resonance spectroscopic imaging in newly diagnosed glioblastoma: predictive value for the site of postradiotherapy relapse in a prospective longitudinal study. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):773-81. doi: 10.1016/j.ijrobp.2007.10.039. PMID 18262090